CLINICAL TRIAL: NCT07366723
Title: The Role of cardIac magNeTic rEsonance in surGical Decision Making in Patients With Severe pRimAry miTral rEgurgitation (the INTEGRATE Study)
Brief Title: The Role of cardIac magNeTic rEsonance in surGical Decision Making in Patients With Severe pRimAry miTral rEgurgitation
Acronym: INTEGRATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: L2-495
Record Dates: First submitted 2025-12-03; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Mitral Valve Prolapse; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Prolapse; Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to a CMR-based strategy (unblinded CMR) or usual care (blinded CMR). A randomization list will be generated using SAS statistical software and will be created by the Biostatistics Unit of Centro Cardiologico Monzino IRCCS, without direct contact with trial participants or involvement in the assessment of study eligibility.
  After randomization, patients will be classified as follows:
  * group A: patients with severe MR, as assessed by TTE, with less than severe MR documented by CMR, undergoing clinical follow-up;
  * group B: patients with severe MR, as quantified by both TTE and CMR, undergoing surgery;
  * group C: patients with severe MR, as assessed by TTE, undergoing surgery as per clinical practice.
  After surgery, baseline CMR of Group C will be unblinded. Then, patients of group C will be furtherly divided into two subgroups: those having less than severe MR as assessed by CMR (subgroup C1) and those with severe MR (subgroup C2).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blinded CMR - Group C1 (Active Comparator): Patients undergoing sugery based on TTE, showing less than severe MR by CMR
  Interventions: Procedure: mitral valve surgery
- Unblinded CMR - Group A (Other): Patients with severe MR, as assessed by TTE, with less than severe MR documented by CMR (Group A), undergo clinical follow-up.
  Interventions: Other: Clinical Follow up
- Unblinded CMR - Group B (Active Comparator): Patients with severe MR, as quantified by both TTE and CMR, undergo surgery.
  Interventions: Procedure: mitral valve surgery
- Blinded CMR - Group C2 (Active Comparator): Patients undergoing surgery based on TTE, showing severe MR by CMR
  Interventions: Procedure: mitral valve surgery

INTERVENTIONS:
Procedure: mitral valve surgery — mitral valve repair or replacement
  Arms: Blinded CMR - Group C1; Blinded CMR - Group C2; Unblinded CMR - Group B
Other: Clinical Follow up — Patients undergo clinical active surveillance.
  Arms: Unblinded CMR - Group A

SUMMARY:
Mitral regurgitation (MR) is the second most frequent valvular heart disease and the second most frequent indication for valve surgery in Europe.

The management of patients with MV prolapse (MVP) and severe MR is mainly guided by symptoms, left ventricular (LV) dimensions and ejection fraction (EF), pulmonary artery systolic pressure (PASP) and atrial fibrillation (AF) occurrence.

According to the ESC/EACTS guidelines, surgical treatment of severe primary MR is indicated (recommendation Class I, Level B) in case of:

* symptomatic patients considered operable by the Heart Team;
* asymptomatic patients with LV dysfunction, intended as a LVEF ≤ 60% and/or LV end-systolic diameter (LVESD) ≥ 40 mm or LVESD indexed for body mass area (LVESDi) ≥ 20 mm/m2;
* low-risk asymptomatic patients without LV dysfunction (LVEF > 60%, LVESD < 40 mm, LVESDi < 20 mm/m2) when a durable result is likely, if at least 3 of the following criteria are fulfilled:

  * AF secondary to MR;
  * PASP value at rest > 50 mmHg;
  * significant left atrium (LA) dilation, intended as LA volume index ≥ 60 mL/m2 or diameter ≥ 55 mm
  * concomitant secondary tricuspid regurgitation ≥ moderate.

Surgery should be considered (recommendation Class IIa, Level B) in asymptomatic patients with preserved LV function (LVEF > 60%, LVESD < 40 mm, LVESDi < 20 mm/m2), when one of the following findings is present1:

* AF secondary to MR;
* PASP value at rest > 50 mmHg;
* LA volume index ≥ 60 mL/m2 or diameter ≥ 55 mm, provided surgical risk is low, surgery is performed in a Heart Valve Center and a durable MV repair is likely.

Preliminary data suggest that in patients with MVP, especially with Barlow's disease phenotype, left-sided chambers' enlargement and functional impairment may be disproportionate related to MR grade. Indeed, patients with BD and ≤ mild-to-moderate MR show larger LA and LV dimensions as compared to controls matched for age, gender and cardiovascular risk factors. These findings challenge the assumption that LA and LV remodeling is a direct effect of volume overload, with possible implications regarding the indication for MV intervention.

On the other hand, low mortality and good durability of valve repair has led some experienced centers to perform also early surgery, namely in any asymptomatic patient with severe MR, normal LV size and function, regular sinus rhythm, normal PASP and normal LA size, as long as surgical risk is very low and likelihood of successful valve repair is high. However, some studies have demonstrated that asymptomatic patients with severe degenerative MR can be safely followed up in experienced hands and remain free of indications for surgery for extensive periods of time. A watchful waiting strategy resulted in timely referral to surgery, excellent long-term survival, and good surgical outcomes, though requiring careful and active surveillance. Several authors agree that prospective randomized trials comparing active surveillance and early elective surgery are needed. There are also data suggesting that MR quantification by CMR has better discriminative power in identifying asymptomatic patients with degenerative MR and adverse outcomes as compared to the echocardiographic-derived integrative approach. Further prospective studies are necessary to validate these preliminary findings.

DETAILED DESCRIPTION:
The present study is a multicenter, prospective, interventional, open randomized controlled trial. Patients will be screened for study eligibility by the clinical research staff of each investigational site. Patients meeting all inclusion criteria will be asked to sign an informed consent document prior to any trial-specific examinations and/or procedures, provided they do not have any of the exclusion criteria. After signing the informed consent, a structured interview will be performed and a clinical history obtained, assessing the presence of common cardiac risk factors, symptoms, and drug therapy (with a specific focus on anti-remodeling drugs, such as angiotensin-converting enzyme inhibitors/angiotensin II receptor blockers and mineralocorticoid receptor blockers). A Quality of Life (QoL) questionnaire will be administered13. Physical examination, rest ECG, CMR and a cardiopulmonary exercise test (CPET) will be also performed.

Subjects will be assigned a subject number upon enrolment. Afterwards, they will be randomized in a 1:1 ratio to a CMR-based strategy (unblinded CMR) or usual care1 (blinded CMR).

A randomization list will be generated using SAS statistical software (version 9.4, SAS Institute, Cary, NC, USA) and will be created by the Biostatistics Unit of Centro Cardiologico Monzino IRCCS, without direct contact with trial participants or involvement in the assessment of study eligibility.

After randomization, patients will be classified as follows (Figure 1 and 2):

* group A: patients with severe MR, as assessed by TTE, with less than severe MR documented by CMR, undergoing clinical follow-up;
* group B: patients with severe MR, as quantified by both TTE and CMR, undergoing surgery;
* group C: patients with severe MR, as assessed by TTE, undergoing surgery as per clinical practice.

After patients of group B and C have undergone surgery, baseline CMR of Group C will be unblinded. Then, patients of group C will be furtherly divided into two subgroups: those having less than severe MR as assessed by CMR (subgroup C1) and those having severe MR (subgroup C2).

At 1-year and 2-year follow-up after enrolment (group A) and after surgery (groups B and C), all patients will undergo a complete evaluation including a clinical interview and physical examination, administration of QoL questionnaires, performance of TTE, CMR and CPET.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* patients agree to all provisions of the protocol;
* patient can give informed consent;
* TTE diagnosis of MVP (defined as a systolic displacement of one or both mitral leaflets ≥ 2 mm above the plane of the MV annulus in long-axis views), and chronic severe MR;
* no symptoms;
* LVEF > 60%, LVESD < 40 mm and LVESDi < 20 mm/m2;
* sinus rhythm;
* PASP value at rest < 50 mmHg;
* LA volume index ≥ 60 mL/m2 or diameter ≥ 55 mm or normal LA size if likelihood of a successful and durable repair without residual MR is >95% and expected mortality rate is <1%
* ongoing adequate treatment per applicable standards;
* patient referred for isolated MV repair or replacement;
* willingness to undergo TTE, CMR and CPET at different timepoints

Exclusion Criteria:

* inability to provide informed consent;
* pregnancy or planned pregnancy within next 2 years;
* poor TTE image quality;
* usual contraindications to CMR and/or to gadolinium administration;
* inability to sustain a breath hold;
* known intracardiac shunts;
* coexistence of other cardiomyopathies or other > mild valve diseases;
* untreated clinically significant coronary artery disease requiring revascularization;
* planned concomitant cardiac surgical procedures (e.g. other valve procedures, or coronary artery bypass);
* need for an emergent/urgent surgery for any reason or any planned cardiac surgery within the next months;
* hemodynamic instability requiring inotropic support or mechanical heart assistance;
* sustained cardiac arrhythmias;
* active endocarditis;
* like expectancy < 12 months due to non-cardiac conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of adverse and reverse LV remodeling | up to 24 months
  The primary efficacy aim is to demonstrate that in patients managed based on CMR results ("unblinded CMR") the proportion of inappropriate clinical decisions is lower as compared to the proportion of inappropriate clinical decisions in patients managed on the basis of TTE results ("blinded CMR").
  In group A:
  * clinical decision will be considered appropriate in case reverse LV remodeling, or no LV remodeling is observed by CMR at 2-year follow-up
  * clinical decision will be considered inappropriate in case adverse LV remodeling by CMR occurs at 2-year follow-up.
  In groups B and C:
  * clinical decision will be considered appropriate in case reverse LV remodeling by CMR occurs at 2-year follow-up
  * clinical decision will be considered inappropriate in case adverse LV remodeling, or no LV remodeling is observed by CMR at 2-year follow-up.
  Operational definitions:
  Adverse LV remodeling=increase in LV EDV >/= 10% vs baseline. Reverse LV remodeling=reduction in LV EDV >/= 30% vs. baseline.

SECONDARY OUTCOMES:
Rate of composite clinical endpoints | up to 24 months
  To demonstrate that freedom from a composite of
  * hospitalization for heart failure
  * Class I indications for surgery
  * atrial fibrillation documentation
  * PASP > 50 mmHg at TTE in the "unblinded CMR" groups is non inferior to freedom from the same events observed in the "blinded CMR" groups at 2-year follow-up, by more than a clinically relevant margin (at most 3%).
  Heart failure hospitalization is defined as an event meeting the following criteria:
  * subject has clinical signs and/or symptoms of heart failure, requires hospitalization in the hospital for at least 24h, and requires intravenous or invasive treatment for heart failure;
  * subject arrives in the emergency department with clinical presentation meeting the criteria of heart failure but dies in the emergency department before hospital admission.
rate of mortality | up to 24 months
  To demonstrate that freedom from cardiovascular death at 2-year follow-up in Groups A+B is non inferior to freedom from the same event in Groups C1+C2.
  Operational definitions: cardiovascular death at 2-year follow-up is intended as any one of the following: any death due to cardiac cause (e.g. myocardial infarction, worsening heart failure); unwitnessed death and death of unknown cause; death caused by non-coronary vascular conditions such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, or other vascular disease.
Measure of exercise capacity | up to 24 moths
  To demonstrate that exercise capacity at 2-year follow-up, as assessed by CPET parameters (peak VO2), is non inferior in the "unblinded CMR" groups as compared to "blinded CMR" groups.
SF-36 Health Survey questionnaire | up to 24 months
  To demonstrate that quality of life at 2-year follow-up, as assessed by the SF-36 Health Survey questionnaire, (from 0 to 100 which is best condition ) is non inferior in the "unblinded CMR" groups as compared to "blinded CMR" groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Pontone, MD, Principal Investigator — Centro Cardiologico Monzino, IRCCS Milan 20131
Locations (1):
- Centro Cardiologico Monzino, IRCCS, Milan, MI, Italy